CLINICAL TRIAL: NCT05320302
Title: Interventional, Open-Label, Positron Emission Tomography (PET) Study With [11C]-Lu AF88370 Investigating Blood-Brain Barrier Penetration of Lu AF88370 in Healthy Men
Brief Title: A Brain Imaging PET Study of [11C]-Lu AF88370 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19874A; 2021-005082-40 (EudraCT Number)
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]-Lu AF88370 (Experimental): Participants will receive [11C]-Lu AF88370 via an intravenous cannula on Day 1.
  Interventions: Drug: [11C]-Lu AF88370

INTERVENTIONS:
Drug: [11C]-Lu AF88370 — PET ligand in a single intravenous bolus injection

SUMMARY:
The main goals of the study are to assess uptake and distribution of Lu AF88370 in the brain when given at tracer levels (microdose) in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30.0 kilograms (kg)/square meter (m^2) at the Screening Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical and neurological examination, vital signs, an ECG, and the results of the clinical chemistry, hematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the first dose of study drug or <5 half-lives prior to the Screening Visit for any medication taken.
* The participant has received a COVID-19 vaccination within the last 30 days before receiving first dose of study drug.
* The participant has had surgery or trauma with significant blood loss <6 months prior to the first dose of the study drug.
* The participant is exposed to significant levels of ionising radiation at work.

Note: Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Whole Brain Total Distribution Volume (VT) of [11C]-Lu AF88370 | Day 1
VT of [11C]-Lu AF88370 in Regions of Interest (ROI) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Invicro, London, United Kingdom